CLINICAL TRIAL: NCT01376128
Title: Special Drug Use Investigation for PAXIL Tablet (Pediatric Panic Disorder)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112309
Record Dates: First submitted 2011-06-09; First posted 2011-06-20 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Paroxetine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed PAXIL: Pediatric subjects with panic disorder prescribed PAXIL during study period
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Paroxetine

SUMMARY:
The objectives of this survey was to retrospectively collect and evaluate the information on the efficacy and safety of PAXIL tablets ("PAXIL", hereinafter) in pediatric subjects (aged under 18) with panic disorder under conditions of actual use.

ELIGIBILITY:
Inclusion Criteria:

* Aged under 18 at the time of the panic disorder diagnosis
* Aged under 18 on the starting day of PAXIL treatment
* Having been making periodic visits to the hospital to receive treatment for panic disorder

Exclusion Criteria:

* Subjects who have been treated with paroxetine prior to this investigation
* Subjects with hypersensitivity to paroxetine
* Subjects taking monoamine oxidase inhibitors (MAOIs) or within 2 weeks of stopping treatment with MAOIs
* Concomitant use in patients taking pimozide

Max Age: 17 Years | Sex: All
Age Groups: Child
Study Population: Male and female Japanese subjects whose age is under 18 with panic disorder, who are considered appropriate to prescribe paroxetine tablet according to the prescribing information
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events in Japanese pediatric subjects with panic disorder treated with paroxetine tablet based on prescribing information under the conditions of general clinical practice | From the starting day of the treatment to the time of treatment termination/discontinuation was assessed from 1 month at minimum up to 2 years
Efficacy evaluation based on overall improvement | From the starting day of the treatment to the time of treatment termination/discontinuation was assessed from 1 month at minimum up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline